CLINICAL TRIAL: NCT06092281
Title: Effect of Questionnaires and Feedback on the Patient Compliance for Endoscopic Surveillance After Endoscopic Submucosal Dissection: a Prospective, Randomized Controlled, Superiority Trial.
Brief Title: Effect of Questionnaires and Feedback on the Patient Compliance for Endoscopic Surveillance After ESD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20232292-F-1
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Patient Compliance
Keywords: compliance; endoscopic submucosal dissection; surveillance; post-ESD
MeSH Terms: conditions — Patient Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Experimental): Patients after ESD are informed on follow-up instructions by doctors about the follow-up requirements before discharge, and complete a questionnaire without compliance-related education.
  Interventions: Behavioral: Questionnaire without compliance-related education
- Questionnaire Arm (Experimental): In addition to receiving the same follow-up instructions as the control group, patients need to complete a questionnaire on compliance-related education before discharge. Based on the responses, nurses provide feedback and guidance.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Patients after ESD need to complete a questionnaire on compliance-related education before discharge. The questionnaire includes the following information:
  1. General information about the patient (e.g., education level, place of residence, economic status, employment status, family history of neoplasms, whether the patient or immediate family member has a medical background, number of previous endoscopic examinations, etc.)
  2. Awareness of follow-up examinations (e.g., knowledge about the timing of the first follow-up, the process of follow-up examinations, related educational issues about follow-up, etc.)
  3. Awareness of the disease (self-perceived tumor is benign or malignant, whether lifestyle changes are required, etc.)
  Arms: Questionnaire Arm
Behavioral: Questionnaire without compliance-related education — Patients after ESD need to complete a questionnaire without compliance-related education before discharge. The questionnaire includes only general information about the patient (e.g., education level, place of residence, economic status, employment status, family history of neoplasms, whether the patient or immediate family member has a medical background, number of previous endoscopic examinations, etc.)
  Arms: Control Arm

SUMMARY:
Endoscopic submucosal dissection (ESD) is now considered the standard treatment for early gastrointestinal neoplasms. However, there is still a possibility of developing local recurrence or metachronous neoplasia after ESD. Regular endoscopic surveillance after ESD can identify and remove local recurrences and metachronous lesions early, improving patient prognosis. However, the patient compliance with post-ESD endoscopic surveillance is currently unclear, and many patients fail to adhere to the scheduled follow-up. A prospective, randomized controlled, superiority trial was designed to evaluate whether completing a questionnaire and receiving feedback on compliance-related education can improve patient compliance with post-ESD endoscopic surveillance, in comparison to those who did not complete the compliance-related education questionnaire. Additionally, the investigators intend to investigate the factors that influence patient compliance.

This study will consist of two parts.

Part 1 will assess whether the completion of questionnaire and feedback on compliance-related education can improve short-term patient compliance with post-ESD endoscopic surveillance, and investigate factors influencing short-term patient compliance.

Part 2 will assess whether the completion of questionnaire and feedback on compliance-related education can improve long-term patient compliance with post-ESD endoscopic surveillance, and investigate factors influencing patient compliance.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled, superiority trial. The study population consists of patients after ESD for mucosal lesions at Xijing Hospital. In the control arm, patients after ESD are informed on follow-up instructions by doctors about the follow-up requirements before discharge, and complete a questionnaire without compliance-related education. In the questionnaire arm, in addition to receiving the same follow-up instructions as the control arm, patients need to complete a questionnaire on compliance-related education before discharge. Based on the responses, nurses provide feedback and guidance. Patients and doctors will be blind to the group of patients during the trial process. Our objective is to evaluate whether completing a questionnaire and receiving feedback on compliance-related education can improve patient compliance with post-ESD endoscopic surveillance, in comparison to those who did not complete the compliance-related education questionnaire. Additionally, the investigators intend to investigate the factors that influence patient compliance.

Part 1 will assess whether the completion of questionnaire and feedback on compliance-related education can improve short-term patient compliance with post-ESD endoscopic surveillance, and investigate factors influencing short-term patient compliance. Part 1 will be expected to include 220 post-ESD patients randomized 1:1 into the questionnaire arm and control arm. Sample size calculation is based on short-term compliance data from a pilot trial, with a 20% difference between the two groups. Under the conditions of an α error of 5% (in a one-sided test) and power of 80%, assuming a superiority margin of 5%, a sample size of 220 cases is required.

Part 2 will assess whether the completion of questionnaire and feedback on compliance-related education can improve long-term patient compliance with post-ESD endoscopic surveillance, and investigate factors influencing patient compliance. Part 2 will be expected to include 500 post-ESD patients randomized 1:1 into the questionnaire arm and control arm. Under the conditions of an α error of 5% (in a one-sided test) and power of 80%, assuming a 20% difference between the two groups in long-term compliance outcome, a superiority margin of 10%, and rounding up, a sample size of 500 cases is required.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) after ESD for mucosal lesions.

Exclusion Criteria:

* Patients after ESD for submucosal tumors, e.g. stromal tumors, neuroendocrine tumors;
* Additional radical surgery after ESD procedure;
* Past history of ESD procedure or local recurrence;
* Severe comorbidities with a life expectancy of <6 months as judged by the investigator;
* Unable to cooperate with information collection due to mental disorders, severe neurosis, or dysgnosia;
* Unable to understand or unwilling to sign a written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: short-term endoscopic surveillance compliance | From enrollment to the end of the first endoscopic surveillance (3 months)
  Patients who undergo their first endoscopic surveillance within 3 months after ESD are considered to have good compliance, otherwise they are considered to have poor compliance.
Part 2: long-term endoscopic surveillance compliance | From enrollment to the end of the last endoscopic surveillance (1-5 years)
  The criteria for endoscopic surveillance after ESD in this study are as follows: (1) For patients with non-neoplastic lesions and benign tumors after ESD, a follow-up of at least 1 year is required; (2) For patients with low-grade intraepithelial neoplasia and adenoma after ESD, a follow-up of at least 1 year is required; (3) For patients with high-grade intraepithelial neoplasia, a follow-up of at least 3 years is required, with an interval not exceeding 2 years; (4) For patients with carcinoma, a follow-up of at least 5 years is required, with an interval not exceeding 2 years. The criteria for assessing the compliance of endoscopic surveillance in this study are as follows: Patients who undergo endoscopic surveillance according to the above-mentioned criteria are considered to have good compliance, otherwise they are considered to have poor compliance.

SECONDARY OUTCOMES:
Part 1: Ulcer scar rate | From enrollment to the end of the first endoscopic surveillance (3 months)
  Percentage of people with ulcer scar stage at first endoscopic surveillance after ESD. The investigators will evaluate ulcer scar rates using a gastric ulcer staging system and measure the ulcer size.
Part 1: Correlated Factors for short-term endoscopic surveillance compliance | From enrollment to the end of the first endoscopic surveillance (3 months)
  The short-term endoscopic surveillance compliance may be influenced by other factors. Patients who undergo their first endoscopic surveillance within 3 months after ESD are considered to have good compliance, otherwise they are considered to have poor compliance. First, univariate analysis will be used to identify potential factors influencing short-term endoscopic surveillance compliance. Then, all possible factors will be included in multivariate analysis.
Part 2: Incidence of metachronous lesions | Up to 5 years
  Metachronous lesions are defined as lesions diagnosed at a minimum interval of 6 months after the initial neoplasia, and the location and pathological type of the lesion are different from the initial neoplasia.
Part 2: Incidence of local recurrence | Up to 5 years
  Percentage of patients with local recurrence detected during follow-up
Part 2: Overall survival rate | 5 years
  Percentage of people still alive at 5 years after ESD
Part 2: Correlated Factors for long-term endoscopic surveillance compliance | From enrollment to the end of the last endoscopic surveillance (1-5 years)
  The long-term endoscopic surveillance compliance may be influenced by other factors. Patients who undergo endoscopic surveillance according to the above-mentioned criteria (see Outcome 2) are considered to have good compliance, otherwise they are considered to have poor compliance. First, univariate analysis will be used to identify potential factors influencing long-term endoscopic surveillance compliance. Then, all possible factors will be included in multivariate analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, Principal Investigator — Xijing Hospital of Digestive DIsease
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ono H, Yao K, Fujishiro M, Oda I, Uedo N, Nimura S, Yahagi N, Iishi H, Oka M, Ajioka Y, Fujimoto K. Guidelines for endoscopic submucosal dissection and endoscopic mucosal resection for early gastric cancer (second edition). Dig Endosc. 2021 Jan;33(1):4-20. doi: 10.1111/den.13883. Epub 2020 Dec 9. PMID 33107115
- [Background] Tanaka S, Kashida H, Saito Y, Yahagi N, Yamano H, Saito S, Hisabe T, Yao T, Watanabe M, Yoshida M, Saitoh Y, Tsuruta O, Sugihara KI, Igarashi M, Toyonaga T, Ajioka Y, Kusunoki M, Koike K, Fujimoto K, Tajiri H. Japan Gastroenterological Endoscopy Society guidelines for colorectal endoscopic submucosal dissection/endoscopic mucosal resection. Dig Endosc. 2020 Jan;32(2):219-239. doi: 10.1111/den.13545. Epub 2019 Dec 27. PMID 31566804
- [Background] Ishihara R, Arima M, Iizuka T, Oyama T, Katada C, Kato M, Goda K, Goto O, Tanaka K, Yano T, Yoshinaga S, Muto M, Kawakubo H, Fujishiro M, Yoshida M, Fujimoto K, Tajiri H, Inoue H; Japan Gastroenterological Endoscopy Society Guidelines Committee of ESD/EMR for Esophageal Cancer. Endoscopic submucosal dissection/endoscopic mucosal resection guidelines for esophageal cancer. Dig Endosc. 2020 May;32(4):452-493. doi: 10.1111/den.13654. PMID 32072683
- [Background] Pimentel-Nunes P, Libanio D, Bastiaansen BAJ, Bhandari P, Bisschops R, Bourke MJ, Esposito G, Lemmers A, Maselli R, Messmann H, Pech O, Pioche M, Vieth M, Weusten BLAM, van Hooft JE, Deprez PH, Dinis-Ribeiro M. Endoscopic submucosal dissection for superficial gastrointestinal lesions: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2022. Endoscopy. 2022 Jun;54(6):591-622. doi: 10.1055/a-1811-7025. Epub 2022 May 6. PMID 35523224